CLINICAL TRIAL: NCT03656328
Title: Supplementation With Lacobacillus Reuteri ATCC PTA 4659 in Patients Affected by Acute Uncomplicated Diverticulitis : a Randomized Double-blind Placebo Controlled Trial
Brief Title: Supplementation With Lacobacillus Reuteri ATCC PTA 4659 in Patients Affected by Acute Uncomplicated Diverticulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, OJETTI VERONICA, Adjuct Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1398
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Acute Diverticulitis
Keywords: probiotics; inflammation markers

STUDY DESIGN:
Intervention Model Description: double blind
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactobacillus Reuteri 4659 (Experimental): This Arm received standard antibiotic therapy, consisting of ciprofloxacin 400 mg twice a day and metronidazole 500 mg three times a day for seven days, with supplementation with the probiotic L. reuteri 4659 twice a day for 10 days
  Interventions: Dietary Supplement: Lactobacillus Reuteri 4659
- Placebo (Placebo Comparator): This arm received the same standard antibiotic therapy and a matching placebo for the same periods.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus Reuteri 4659 — supplementation with L. reuteri 4659 twice a day for 10 days during the standard antibiotic therapy
  Arms: Lactobacillus Reuteri 4659
Dietary Supplement: Placebo — supplementation with a Placebo capsule twice a day for 10 days during the standard antibiotic therapy
  Arms: Placebo

SUMMARY:
Acute Uncomplicated Diverticulitis (AUD) is defined as inflammation of the colon diverticulum, often involving the colic wall and pericolic fat. In a double-blind RCT study, the investigators tested the efficacy of Lactobacillus reuteri ATCC PTA 4659 (L. reuteri), a specific strain with anti-inflammatory effect in association with conventional antibiotics, in treating AUD, compared with conventional antibiotic therapy plus placebo. A primary outcome was reduced abdominal pain and inflammatory markers (C-RP) in the group treated with L. reuteri compared with the placebo. A secondary outcome was reduced hours of hospitalization in the L. reuteri group.

A double-blind, placebo RCT was conducted with 90 consecutive patients with a diagnosis of AUD treated at the Emergency Department of Foundation Poli-clinico A. Gemelli Hospital. Following a routine blood test and determination of C-reactive protein (C-RP) value, all patients were admitted to the Brief Observation Unit (BOU) and randomly as-signed to two groups:

* Group A : Treated with ciprofloxacin 400 mg twice a day and metronidazole 500 mg three times a day for one week, plus supplementation with L. reuteri twice a day for 10 days.
* Group B : Treated with the same antibiotic therapy as Group A for one week, plus placebo twice a day for 10 days.

All patients completed a daily Visual Analog Scale (VAS) for abdominal pain, with a range from 0 (asymptomatic) to 10. C-RP value was determined again at 72 hours.

DETAILED DESCRIPTION:
Patients are evaluated in a clinical setting by a physician at enrolment in the study, every day during hospitalization, and at the end of therapy. At enrolment, a medical history review (including drugs taken), physical examination, laboratory tests (blood cell count, hepatic and renal function, electrolytes, C-RP) and abdominal CT scan were performed.

All patients presented with AUD (Hinchey classification grade 0). All patients were given a Visual Analog Scale (VAS) ranging from 0 to 10, where 0 is asymptomatic and 10 is the worst pain they could have, to complete during the 10 days of the study.

Patients were also asked to complete a diary, in order to record any 'adverse experience' (causing discomfort and/or interrupting the subject's usual activity) during the treatment periods, and to record every time they did not consume the prescribed doses. The diary was analyzed by physicians.

The patients are randomly assigned into two groups, according to an automatically generated randomization list in a 1:1 ratio, using statistical software:

Group A received standard antibiotic therapy, consisting of ciprofloxacin 400 mg twice a day and metronidazole 500 mg three times a day for seven days, with supplementation with the probiotic L. reuteri 4659 twice a day for 10 days.

Group B received the same standard antibiotic therapy as group A and a matching placebo for the same periods.

Patients were informed by an investigator (blind) that such a supplement could help in improving the inflammation associated with diverticulitis. Boxes containing placebo had the same shape dimensions, and trade mark indication and contained the same amount of capsules as L. reuteri boxes, and they were provided by the same probiotic producer.

The supplement of L. reuteri 4659 was administered in a dose of 108 colony-forming units (CFU), in capsules 30 minutes after food. During the study period, patients were instructed to store the product according to the recommended temperature. In particular, the capsules could be stored at room temperature (25°C). Because L. reuteri is a living organism, over long storage periods it is preferable not to freeze the capsules, but to refrigerate them at 2-8°C.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* No reported allergies to contrast agents or antibiotics
* Informed consent
* Diagnosis of AUD confirmed by abdomen CT scan

Exclusion Criteria:

* <18 years
* Pregnancy or breastfeeding
* Concomitant or recent (7-10 days) participation in another clinical trial
* Concomitant or recent (7-15 days) intake of probiotics or antibiotics
* Major concurrent diseases (hepatological, renal, tumor)
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis) or other organic gastrointestinal disease
* Allergies to contrast agents or antibiotics
* Mental illness or inability to adhere to protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
reduction of abdominal pain | 10 days
  evaluation with a Visual Analog Scale of abdominal pain between the two arms. The Visual Analog Scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured, like pain. it goes from 0 (asymptomatic) to 10 (the maximum pain).

SECONDARY OUTCOMES:
reduction of inflammatory markers | 72 hours
  evaluation of C-reactive Protein at enrollment and after 72 hours of therapy
comparisons of hours of hospitalization | 5 days
  comparison of hospitalization time between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Ojetti, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Policlinico universitario agostino gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petruzziello C, Migneco A, Cardone S, Covino M, Saviano A, Franceschi F, Ojetti V. Supplementation with Lactobacillus reuteri ATCC PTA 4659 in patients affected by acute uncomplicated diverticulitis: a randomized double-blind placebo controlled trial. Int J Colorectal Dis. 2019 Jun;34(6):1087-1094. doi: 10.1007/s00384-019-03295-1. Epub 2019 Apr 22. PMID 31011868